CLINICAL TRIAL: NCT04511494
Title: Oral Immunotherapy for Young Children With Peanut Allergy - Small Children OIT (SmaChO)
Brief Title: Oral Immunotherapy for Young Children With Peanut Allergy - Small Children OIT
Acronym: SmaChO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Stockholm South General Hospital (Other)
Responsible Party: Principal Investigator, Carina Uhl, PhD student, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-04645
Record Dates: First submitted 2020-05-11; First posted 2020-08-13 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Peanut Allergy
Keywords: Peanut Hypersensitivity; Immunotherapy; Child preschool; Arachis
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Blinded randomisation process after a positive baseline peanut challenge (for both participants, care provider and investigator) by opaque envelops.
  After the child is randomised to treatment or avoidance, everyone (particpant, care provider and investigator) know if the child is in the treatment or avoidance group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- OIT peanut (Active Comparator): Children with peanut allergy receiving peanut OIT. Peanut challenge are done before randomization and one and three years after inclusion.
  n=50 patients
  Interventions: Dietary Supplement: Peanut (bamba)
- Peanut avoidance (No Intervention): Children with peanut allergy not undergoing OIT peanut. Peanut challenge are done Before randomization and one and three years after inclusion.
  n=25 patients
- Healthy controls (No Intervention): Control Group with non-allergic, age-matched children. No challenges are performed in this group.
  n=30 patients
- Children not reacting at the baseline peanut challenge (No Intervention): Peanut-allergic children not reacting at the baseline peanut challenge, will not be eligible for randomisation. They will have a clinical visit after 1+3 years. No more challenges in this group.
  n=X patients

INTERVENTIONS:
Dietary Supplement: Peanut (bamba) — OIT peanut with slow-updosing for 40-60 weeks followed by maintenance. 3 years treatment.
  Arms: OIT peanut

SUMMARY:
Open label study with peanut oral immunotherapy (OIT). Peanut allergic children aged 1-3 years of age will be randomized 2:1 to:

1. Peanut OIT with slow up-dosing (40-60 weeks) up to a maintenance dose of 285 mg daily oral peanut protein or
2. Control group with peanut allergic children who do not undergo OIT.
3. In addition, a group of healthy children without allergic diseases will be included in the study.

The primary outcome is tolerance to at least 750 mg peanut protein at a challenge after 3 years and sustained unresponsiveness (i.e. tolerance) to 750 mg peanut protein after 3 years of OIT followed by 4-6 weeks of avoidance.

Efficacy and safety will be compared between group 1 and 2. Group 3 is a control group for analyses of immunological markers.

DETAILED DESCRIPTION:
Problem: Today there is no clinically available treatment for peanut allergy. Oral Immunotherapy (OIT) studies have shown promising results, particularly in younger children (<4 years).

Intervention: Peanut OIT in children aged 1-3 years with peanut allergy (clinical symptoms at peanut challenge and IgE >0.1 kU /l to peanut and/or Ara h 2).

Comparison: Three groups are compared. Peanut allergic children are randomized 2:1 to group 1 (active OIT) or group 2 (control). Group 3 consists of age-matched non-allergic children:

Group 1; Children with peanut allergy receiving peanut OIT, slow up-dosing, 40-60 weeks, until the maintenance dose 285 mg peanut protein. Three years' treatment. (n=50 patients)

Group 2; Age-matched children with peanut allergy who do not undergo OIT peanut (peanut avoidance group). Peanut challenges are performed one and three years after inclusion. (n=25 patients)

Group 3; Healthy, non-allergic, age-matched children. No challenges are performed in this group. (n=30 patients)

Group 4; Children not reacting at the baseline peanut challenge (n=9 patients)

Inclusion of study subjects: A review of samples sent to the Karolinska University Laboratory for IgE-ab responses to peanut/Ara h 2 for children in the Stockholm area aged 1-3 years is used for identification of potential participants to whom a letter is sent with information about the study. The families are randomized 2:1 to OIT or control group, group 1 or group 2.

Children without allergies, healthy controls (group 3), will be included from Västerås Hospital.

If children are included in the study but they do not not react at the baseline peanutchallenge, they will not have any intervention (are not eligible to randomisation) and will have a follow-up after 1+3 years (without peanut challenges), group 4.

Outcomes: The primary outcome is defined as sustained unresponsiveness to 750 mg peanut protein (cumulative dose) at an open oral peanut challenge after 3 years of OIT followed by 4-6 weeks of avoidance (group 1 and 2).

Secondary outcomes are adverse events among peanut allergic children with/without OIT treatment (group 1 and 2), and changes in quality of life parameters and immunological markers (group, 1, 2, 3).

ELIGIBILITY:
Inclusion Criteria:

* Children 1 - 3 years old at inclusion
* Positive baseline challenge at a maximum of the 250 mg peanut protein-dose with at least one objective symptom, or positive peanut challenge performed in the clinic in a similar way within 1 year from study start.
* IgE-ab to peanut and/or Ara h 2 ≥0.1 kUA/l, analyzed within 12 months from start of study
* Written consent for participation in the study from both Guardians

Exclusion Criteria:

* Other serious illness
* Previously life-threatening anaphylaxis (intensive care), regardless of the triggering agent
* A history of eosinophilic esophagitis (EoE), other eosinophilic gastrointestinal disease, severe chronic gastroesophageal reflux disease (GERD), symptoms of dysphagia, unclear recurrent GI disorders
* Participation in another intervention study, if included in intervention Group
* Severe uncontrolled asthma
* Ongoing medication with biological drugs or oral steroids

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Sustained unresponsiveness to 750 mg peanut protein | 3 years and 4-6 weeks
  Sustained unresponsiveness to 750 mg peanut protein (cumulative dose) at a peanut challenge after 3 years of OIT and 4-6 weeks of peanut avoidance. Measured at a peanut challenge

SECONDARY OUTCOMES:
Adverse events during OIT treatment | 3 years
  Adverse events among peanut allergic children with OIT treatment
Quality of Life Before, during and after OIT peanut | 3 years
  Examine how quality of life, measured with Food Allergy Quality of Life Questionnaire-parental Form (FAQLQ-PF), is affected in families with peanut allergic children undergoing peanut OIT compared to those without peanut OIT. FAQLQ-PF has questions for food-allergy specific QoL with general emotional impact; food anxiety; social and dietary limitations. The FAQLQ-PF has a seven-point scale ranging from 0 (no impact on HRQL) to 6 (extreme impact on HRQL).Overall and domain-specific HRQL scores will be calculated. Higher scores mean a worse outcome and a score of ≥ ±0.5 will be considered clinically relevant.
Intestinal microbiome | 3 years
  The gut microbiome will be investigated with sequencing-based methods to monitor possible changes in the gut microbiota composition and function related to OIT treatment. This will be compared to samples from the non-allergic individuals (reference).
Immunological biomarkers | 3 years
  To study differerent immunological biomarkers (e.g. T-helper cell-population and polarization and IgE levels) before, during and after OIT treatment and compare this to healthy controls. Immunological marker in mononuclear cells in peripheral blood will be analyzed ex vivo with flowcytometri and RNA-sequensingplatforms. Cirkulating immunological factors, e.g. cytokines and chemocines will be analyzed in plasma with ELISA-based methods.Mononuclear cellpopulations in periferal blood will be exposed to different stimuli (such as peanut, anti-C D3/C D28) in vitro, type anf level of reaction in the different cellpopulations will be monitored at mRNA- och protein-level.
Tolerance to peanut protein at a challenge after 3 years | 3 years
  Is OIT peanut with a low dose and slow up dosing strategy in young peanut allergic Children safe and effective? Measured at a peanut challenge
Tolerance to peanut protein at a challenge after 1 year | 1 year
  Is OIT peanut with a low dose and slow up dosing strategy in young peanut allergic children safe and effective? Measured at a peanut challenge

CONTACTS AND LOCATIONS:
Overall Officials: Anna Asarnoj, Principal Investigator — Karolinska Institutet
Locations (1):
- Forskningsenheten Södersjukhuset, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No